CLINICAL TRIAL: NCT02885493
Title: The Elderly 's Parkinsonian March : Risk Estimation Multiple Drops From an Evaluation Grid Covering the March, Executive Functions, Vision and Anxiety.
Brief Title: Evaluation of Dysfunction of the Basal Ganglia Before a Parkinsonian Walking in the Elderly: Risk of Falling and Confusional State
Acronym: EVAMARAGEX
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5955
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: the Elderly
Keywords: Parkinson march

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Falls is <or = 1 year: Patients whose number of falls is <or = 1 year
  Interventions: Behavioral: tests
- falls is> 1 year: Patients whose numbers falls is> 1 year
  Interventions: Behavioral: tests

INTERVENTIONS:
Behavioral: tests

SUMMARY:
The strong relationship between falling and severity of cognitive impairment in the elderly is well established. The association premorbid gait and executive disorders suggests that they are under tension by the same mechanisms. The gait fortiori neurological are fall risk factors. Dysfunctions underlying disorders as Parkinson called march executive disorders are subcortical origin involving so the basal ganglia. This study is indeed based on the assumption that the dysfunction of the basal ganglia as observed in parkinsonian syndromes resulting in disorders of posture and walking, by dysexecutive syndrome, anxiety and the contrast vision disorders. These gait exposed to falls and dysexecutive these disorders with cognitive impairment and greater susceptibility to confusional states. The executive disorders, gait disorders, anxiety, disturbances of vision and especially saccadic eye movements, impaired vision contrasts are well established in the degenerative parkinsonian syndromes. This study proposes a new approach to assessing gait disorders to define a high risk of falling in the presence of parkinsonian walking in the elderly over 75 years.

ELIGIBILITY:
Inclusion Criteria:

* Age: 75 years,
* man or woman,
* Diagnostic Criteria for Parkinson walking: at least 3 of the following symptoms:
* Loss of swinging arms,
* Decrease in stride walking slowly,
* feet as glued to the ground,
* Trample,
* piece U-turn,
* kyphotic Attitude,
* Tolerance screw physiotherapy screws

Exclusion Criteria:

* Unrecovered delirium,
* Unable to walk for a distance of 6 meters in length without technical assistance,
* Traumatic fall phase of rehabilitation,
* Acute pathology,
* Unstabilized psychiatric pathology,
* Symptomatic orthostatic hypotension,
* Severe depressive syndrome untreated
* Subjects with a sufficient gap to explain the falls:

  * cerebellar syndrome,
  * a pyramidal syndrome with sequelae pyramidal deficit and cortical stroke
  * peripheral pathology,
  * rheumatic disease,
  * orthopedic pathology,
* Mini Metam State Examination <18,
* Parkinsonism induced by neuroleptics,
* Not cured cancer,
* Psychotropic drugs (benzodiazepines and antipsychotics) with significant sedative effect inducing excessive daytime sleepiness namely psychotropic half long life, and high dose over 2 psychotropic
* Severe heart failure
* Severe respiratory failure,
* Associated diseases and treatments interfering

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: the eldery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
falls risks | number of falls during follow-up of 24 months
  Assess Falls development risk in the presence of parkinsonian walking

SECONDARY OUTCOMES:
number of confusional states | follow-up of 24 months
number of hospitalizations | follow-up of 24 months
mortality | follow-up of 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michèle KIESMANN, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kiesmann M, Martin RE, Sauleau E, Bulubas I, Fleury MC, Perisse J, Kaltenbach G, Schmitt E. Diagnosis of vascular parkinsonism: A new tool for gait hypokinesia occurring in older persons. Parkinsonism Relat Disord. 2023 Apr;109:105360. doi: 10.1016/j.parkreldis.2023.105360. Epub 2023 Mar 8. PMID 36921515
- [Derived] Kiesmann M, Sauleau E, Ewald Martin R, Danan J, Sauer A, Konrad S, Blanc F, Vogel T, Kaltenbach G, Schmitt E. Older Persons Displaying Parkinsonian Gait: Prediction and Explanation of the Recurrent Falling Phenomenon and Its Related Poor Prognosis. Gerontology. 2022;68(12):1402-1414. doi: 10.1159/000521503. Epub 2022 Feb 11. PMID 35152218